CLINICAL TRIAL: NCT05057169
Title: Randomized Trial of COVID-19 Booster Vaccinations (Cobovax Study)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: BJC053
Record Dates: First submitted 2021-09-24; First posted 2021-09-27 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: COVID-19 Vaccination
MeSH Terms: interventions — BNT162 Vaccine; sinovac COVID-19 vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- BNT162b2 third dose after two doses of BNT162b2 (Experimental)
  Interventions: Biological: BNT162b2
- CoronaVac third dose after two doses of BNT162b2 (Experimental)
  Interventions: Biological: CoronaVac
- BNT162b2 third dose after two doses of CoronaVac (Experimental)
  Interventions: Biological: BNT162b2
- CoronaVac third dose after two doses of CoronaVac (Experimental)
  Interventions: Biological: CoronaVac

INTERVENTIONS:
Biological: BNT162b2 — BNT162b2 is a nucleoside-modified mRNA encoding the trimerized SARS-CoV-2 spike glycoprotein. The vaccine is formulated in lipid nanoparticles that increase the efficiency of delivery of the mRNA into cells after intramuscular injection. BNT162b2 encodes the SARS- CoV-2 full-length spike, modified by two proline mutations to lock it in the prefusion conformation and more closely recreate the intact virus with which the elicited virus- neutralizing antibodies interact. mRNA vaccines use the pathogen's genetic code as the vaccine; hence they exploit the host cells to translate the code and generate the target spike protein. The protein then acts as an intracellular antigen to stimulate the immune response of the vaccinated individual. The mRNA is then degraded within days.
  Other Names: Comirnaty
  Arms: BNT162b2 third dose after two doses of BNT162b2; BNT162b2 third dose after two doses of CoronaVac
Biological: CoronaVac — CoronaVac is a Vero cell-based, aluminium hydroxide-adjuvanted, β-propiolactone- inactivated vaccine based on the CZ02 strain. This strain of SARS-CoV-2 was isolated from the bronchoalveolar lavage of a hospitalized patient and is closely related to the 2019-nCoV- BetaCoV Wuhan/WIV04/2019 strain. Each 0.5 ml dose is composed of 3 μg of inactivated SARS-CoV-2 virus. The excipients are aluminium hydroxide, disodium hydrogen phosphate, sodium dihydrogen phosphate, sodium chloride, and water for injection.
  Arms: CoronaVac third dose after two doses of BNT162b2; CoronaVac third dose after two doses of CoronaVac

SUMMARY:
Randomized comparison of 3rd dose with inactivated vaccine (CoronaVac) or mRNA vaccine (Comirnaty) in adults who previously received two doses of CoronaVac (Sinovac) or two doses of BNT162b2 (Comirnaty, BioNTech/Fosun Pharma) at least 6 months earlier.

DETAILED DESCRIPTION:
Background: The accrual of population immunity to COVID-19 could allow life to return to pre- pandemic normality. Immunity can be acquired through natural infections or, preferably, by vaccination. An unprecedented global effort has succeeded in developing a number of COVID-19 vaccines. All vaccines against COVID-19 approved until now have originally been developed as either a single dose or following a homologous two-dose regimen. Inactivated COVID-19 vaccines have shown inferior immunogenicity compared to mRNA vaccines but there are no studies comparing the advantages of alternative booster doses in individuals who have previously received two doses of an inactivated COVID-19 vaccine or two doses of an mRNA vaccine.

Aims and primary objectives: The aims of this study are: (1) to compare the SARS-CoV-2 antibody responses to one dose of BNT162b2 (mRNA vaccine, Fosun/BioNTech) versus one dose of CoronaVac (inactivated vaccine, Sinovac) in individuals who have previously received two doses of COVID-19 vaccination using BNT162b2 (mRNA vaccine, Fosun/BioNTech) or CoronaVac (inactivated vaccine, Sinovac), and (2) to assess the reactogenicity and safety of one booster dose of BNT162b2 and CoronaVac. The specific primary objective of our study is to assess the vaccine (humoral) immunogenicity, proxied by SARS-CoV-2 serum neutralizing antibody titers, of one booster dose of BNT162b2 or CoronaVac at 28 days after the booster dose in individuals who have previously received two doses of a COVID-19 vaccine.

Study design: Randomized open label trial in adults aged 18 years of age or older (at enrolment). The duration of participation for each participant will be 12 months from the administration of the vaccination booster dose. The immune response and reactogenicity of one dose of BNT162b2 or CoronaVac will be investigated in individuals who previously received two doses of COVID-19 vaccine at least 6 months earlier. Participants will be enrolled shortly before receiving the booster dose of BNT162b2 (day 0), with blood collection at days 0, 28, 182 and 365 days after enrolment for analysis of humoral immune responses. A subset of 25% of participants will provide additional blood samples at day 0, 7 and 30 for assessment of cellular immune responses.

Main outcomes: The primary outcome is the vaccine (humoral) immunogenicity measured as SARS- CoV-2 serum neutralizing antibodies, evaluated as the geometric mean titer (GMT) at 28 days after the booster doses. The secondary outcomes include (1) a comparison of SARS-CoV-2 serum neutralizing antibodies as the geometric mean fold rise from baseline to each post-vaccination timepoint (i.e. at days 28, 182 and 365); (2) a comparison of cellular immune responses at day 7 and 30 compared to day 0; (3) descriptive analysis of the reactogenicity and safety profiles of the booster doses.

Target population: Adults aged 18 years or older

Number of subjects planned: 400 participants to be recruited in 2021-22

Study Duration: 12 months, from September 2021 through to March 2023

Potential implications: This study will provide important evidence into the comparative effects of using a dose of mRNA vaccine or inactivated vaccine to boost the immune response in individuals that had previously received two doses of COVID-19 vaccination. This information together with data collected on reactogenicity and safety could inform COVID-19 vaccination policy locally and internationally.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older at enrolment.
* Have received two doses of BNT162b2 OR two doses of CoronaVac, with the most recent dose at least six months prior to enrolment.
* Currently resident and planning to remain resident in Hong Kong during the duration of the study, i.e. for 12 months after enrolment.
* Agreement to refrain from blood donation during the course of the study.
* Willing to provide blood samples for all the required time points.
* The individual or their caregiver have a home phone or cellular or mobile phone for communications purpose.
* Capable of providing informed consent.

Exclusion Criteria:

* A history of laboratory-confirmed or clinically confirmed COVID-19 infection prior to enrolment.
* Have previously already received one or two doses of any COVID-19 vaccines except CoronaVac or BNT162b2, for example but not limited to BBIBP-CorV (inactivated vaccine, Sinopharm), AZD1222 (adenovirus vector-based vaccine, Oxford/AstraZeneca), Sputnik V (adenovirus vector-based vaccine, Gamaleya Research Institute) and Ad26.COV2.S (adenovirus vector-based vaccine, Johnson & Johnson).
* Individuals who report any medical condition, or as determined by a clinician, not suitable to receive mRNA or inactivated COVID-19 vaccines, including but not limited to allergies to the active substance or other ingredients of the vaccine.
* Currently with diagnosed medical conditions related to their immune system.
* Use of medication that impairs immune system in the last 6 months, except topical steroids or short-term oral steroids (course lasting ≤ 14 days).
* Administration of immunoglobulins and/or any blood products within 90 days preceding the planned administration of the study vaccines.
* Pregnancy, lactation or intention to become pregnant in the coming 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-11-18 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Geometric mean titer (GMT) of SARS-CoV-2 serum neutralizing antibodies | 28 days after vaccination
  The primary outcome measure is the vaccine (humoral) immunogenicity at 28 days after the booster dose, measured as geometric mean titer (GMT) of SARS-CoV-2 serum neutralizing antibodies using plaque reduction neutralization test (PRNT).

SECONDARY OUTCOMES:
Geometric mean titer (GMT) of SARS-CoV-2 serum neutralizing antibodies | 182 and 365 days after vaccination
  The GMT of SARS-CoV-2 serum PRNT titers after the booster dose at Days 182 and 365.
Geometric mean fold rise of SARS-CoV-2 serum neutralizing antibodies | Day 28, 49, 182 and 365 after vaccination
  The geometric mean fold rise (GMFR) of SARS-CoV-2 serum neutralizing antibody titers from baseline to each post-vaccination timepoint measured.
T-cell responses to vaccination | 7 and 28 days after vaccination
  Vaccine-specific IFN-γ+CD4+ and IFN-γ+CD8+ T-cell response at Day 7 and 28.
Reactogenicity | 7 days after vaccination or until symptoms resolve
  Incidence of solicited local and systemic adverse events after the booster dose of vaccination.
Hospitalizations from any cause | One year after vaccination
  Incidence of hospitalizations during the year after receipt of the booster dose.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin J Cowling, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Leung NHL, Cheng SMS, Cohen CA, Martin-Sanchez M, Au NYM, Luk LLH, Tsang LCH, Kwan KKH, Chaothai S, Fung LWC, Cheung AWL, Chan KCK, Li JKC, Ng YY, Kaewpreedee P, Jia JZ, Ip DKM, Poon LLM, Leung GM, Peiris JSM, Valkenburg SA, Cowling BJ. Comparative antibody and cell-mediated immune responses, reactogenicity, and efficacy of homologous and heterologous boosting with CoronaVac and BNT162b2 (Cobovax): an open-label, randomised trial. Lancet Microbe. 2023 Sep;4(9):e670-e682. doi: 10.1016/S2666-5247(23)00216-1. Epub 2023 Aug 4. PMID 37549680